CLINICAL TRIAL: NCT00480051
Title: RESynchronisation in Patients With Heart Failure and a Normal QRS Duration
Acronym: RESPOND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heart of England NHS Trust (Other)
Collaborators: Sandwell & West Birmingham Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007CD002.GH
Record Dates: First submitted 2007-05-29; First posted 2007-05-30 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Heart Failure, Congestive
Keywords: Cardiac Failure; Pacemaker; Dyssynchrony; Cardiac Magnetic Resonance; Narrow QRS
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Cardiac Resynchronization Pacing

SUMMARY:
Patients who have heart failure and have electrical evidence of delay in the contraction of the left ventricle on an ECG tracing of the heart are eligible for biventricular pacing. Recent work has suggested that patients with heart failure who do not have electrical evidence of conduction delay (normal QRS) may benefit from biventricular pacing. The reliance on ECGs to determine the presence of dyssynchrony is widespread, although the ECG alone is not 100% sensitive and specific. ECG criteria for de-synchrony in heart failure patients are estimated to pick up only 30% of patients with dyssynchrony, and results in patients missing out on a potentially important treatment advance.

We would like to study patients with heart failure who have normal ventricular activation on their ECGs to see whether we can predict those patients who will respond to biventricular pacing.

DETAILED DESCRIPTION:
AIMS and Objectives A randomised controlled clinical trial

Primary objective

• Improvements in 6-min walking distance

Secondary objectives Determine

1. Symptomatic improvement in quality of life, using the Minnesota Living with Heart Failure questionnaire
2. Change in NT pro-BNP and echocardiographic parameters of LV function
3. Does MRI Dyssynchrony Index (CMR-TSI) predicts responders.
4. Morbidity and Mortality using CARE-HF definitions
5. Packer combined clinical composite score

Study Design A pilot randomised controlled clinical trial 60 patients. The biventricular pacemaker with be optimized for both A-V delay and V-V delay.

Subject Selection Source - Patients attending Good Hope Hospital, Sandwell Hospital Centres involved - 2 Eligible Participants - 60 patients with heart failure and narrow QRS.

Inclusion Criteria Sinus rhythm Symptomatic heart failure - NYHA class III or IV ECG QRS duration less than 120 milliseconds LV ejection fraction of less than 35% on echocardiography using Simpsons technique.

Able to give informed consent

Exclusion Criteria Age below 18 Current or planned pregnancy Patient refusal Ventricular tachycardia or ventricular fibrillation Current or recent (within last 30 days) involvement in other studies Requires implantable cardioverter defibrillator (ICD) according to NICE criteria for implantation (England and Wales)

Definition of clinical response:- 20% improvement in 6 minute walk distance or any improvement from 0

Definition of echocardiographic response:- 15% or greater decrease in left ventricular end systolic volume

Follow up 6 weeks and 6 monthly thereafter. Interim results at 6 months. Analysis of results, echocardiograms, MRI and BNP will be blind Walk distance to be measured by unblinded observer and by pedometer.

Randomisation:

Numbered envelopes will be prepared by sponsor (Heart of England NHS Foundation Trust) and kept from researchers. After informed consent, the patient will be enrolled and the technician will draw the result.

This trial was known as the Birmingham biventricular pacing in patients unselected for dyssynchrony (BIPIDS).

ELIGIBILITY:
Inclusion Criteria:

* Sinus rhythm
* Symptomatic heart failure - NYHA class III or IV
* ECG QRS duration less than 120 milliseconds
* LV ejection fraction of less than 35% on echo
* Able to give informed consent

Exclusion Criteria:

* Age below 18
* Current or planned pregnancy
* Patient refusal
* Ventricular tachycardia or ventricular fibrillation
* Current or recent (within last 30 days) involvement in other studies
* Requires implantable cardioverter defibrillator (ICD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Improvements in 6-min walking distance | 6 months

SECONDARY OUTCOMES:
Symptomatic improvement in quality of life, using the Minnesota Living with Heart Failure questionnaire | 6 months
Change in NT pro-BNP and echocardiographic parameters of LV function | 6 months
Does MRI Dyssynchrony Index (CMR-TSI) predicts responders | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Leyva, MD MB BS, Study Chair — University of Birmingham; Paul W Foley, MB ChB MRCP, Principal Investigator — Heart of England NHS Foundation Trust; Kiran Patel, PhD MRCP, Principal Investigator — Sandwell & West Birmingham Hospitals NHS Trust; Berthold Stegemann, PhD, Principal Investigator — Bakken Research Centre, The Netherlands; Russell EA Smith, FRCP MD, Principal Investigator — University Hospital Birmingham
Locations (2):
- United Kingdom (2):
  - Sandwell Hospital, Birmingham
  - Good Hope Hospital, Sutton Coldfield

REFERENCES:
- [Derived] Foley PW, Patel K, Irwin N, Sanderson JE, Frenneaux MP, Smith RE, Stegemann B, Leyva F. Cardiac resynchronisation therapy in patients with heart failure and a normal QRS duration: the RESPOND study. Heart. 2011 Jul;97(13):1041-7. doi: 10.1136/hrt.2010.208355. Epub 2011 Feb 21. PMID 21339317